CLINICAL TRIAL: NCT06900569
Title: Ashwagandha Supplementation for Recovery From Muscle-damaging Exercise and Sleep Quality
Brief Title: Ashwagandha Supplementation for Prevention of Muscle Damage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024_25_06
Record Dates: First submitted 2025-03-15; First posted 2025-03-28 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Muscle Damage
MeSH Terms: interventions — Ashwagandha

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 600 mg/d placebo for 10 days
  Interventions: Dietary Supplement: Placebo
- Ashwagandha (Experimental): 600 mg/d Ashwagandha
  Interventions: Dietary Supplement: Ashwagandha

INTERVENTIONS:
Dietary Supplement: Ashwagandha — 600 mg/d Ashwagandha
  Arms: Ashwagandha
Dietary Supplement: Placebo — 600 mg/d placebo
  Arms: Placebo

SUMMARY:
Ashwagandha is an herbal supplement that has a wide range of benefits related to exercise when supplemented for about 8-12 weeks. This study aims to investigate whether short-term Ashwagandha supplementation can enhance muscle recovery following exercise by measuring muscle strength recovery, swelling, and soreness in the biceps.

DETAILED DESCRIPTION:
The purpose of the study is to determine the effects of Ashwagandha supplementation on recovery from muscle-damaging exercise. Ten to twenty participants will be randomized to receive Ashwagandha supplementation (600 mg/d) or placebo for 10 days. On day 7, participants will perform a muscle damaging exercise session (six sets of concentric and emphasized eccentric repetitions with the biceps). Before and after exercise and at 24, 48, and 72 hours after exercise, isometric muscle strength, muscle swelling (ultrasound), and muscle soreness will be assessed. The investigators hypothesize the Ashwagandha will alleviate symptoms of muscle damage (swelling and soreness) and enhance strength recovery after a bout of muscle-damaging exercise.

ELIGIBILITY:
Inclusion Criteria: male or female, aged 18-35y

-

Exclusion Criteria:

Conditions that may be affected by exercise (determined by "yes" answers to the "Get Active Questionnaire") Pregnant Breastfeeding

Allergies to:

* Dicalcium Phosphate
* Cellulose
* Vegetable magnesium stearate
* Silica

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-22 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Change in isometric biceps strength measured with a dynamometer (Nm) | 72 hours

SECONDARY OUTCOMES:
Change in muscle thickness measured with ultrasound (cm) | 72 hours
Change in muscle soreness measured with a visual analog scale with scores ranging from 0 (no soreness) to 10 (maximal soreness) | 72 hours
Change in sleep quality with the Pittsburgh Sleep Quality Index with scores ranging from 0 (no sleep problems) to 3 (lowest sleep quality) | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No